CLINICAL TRIAL: NCT01828814
Title: Different Strategies for Preventing Severe Acute Malnutrition in Niger: a Pragmatic Trial
Brief Title: Different Strategies for Preventing Severe Acute Malnutrition in Niger
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: United Nations World Food Programme (WFP) (Other)
Responsible Party: Sponsor
Other Study IDs: Epicentre
Record Dates: First submitted 2013-03-04; First posted 2013-04-11 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Malnutrition
Keywords: pediatrics; Ready-to-use Supplementary Food; corn soy blend; cash transfer; prevention of malnutrition; Niger
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- RUSF (500kcal/day) and cash transfer: Monthly distributions of Ready-to-use Supplementary Food (RUSF) 500kcal per day associated with cash transfer during hunger gap (5 months) then RUSF 500kcal/day for 10 months
- Super Cereal Plus (SC+): Monthly distributions of SC+ 800kcal per day during hunger gaps (5 months twice) and SC+ 400kcal per day in-between (5 months)
- RUSF: Monthly distributions of Ready-to-use Supplementary Food (RUSF) 500kcal per day during hunger gaps (5 months twice) and RUSF 250kcal per day in-between (5 months)
- RUSF (250kcal/day) and cash transfer: Monthly distributions of Ready-to-use Supplementary Food (RUSF) 250kcal per day associated with cash transfer during hunger gap (5 months) then RUSF 250kcal/day for 10 months
- SC+ and cash transfer: Monthly distributions of Super Cereal Plus (SC+) 800 kcal per day associated with cash transfer during hunger gap (5 months)
- SC+ and household ration: Monthly distributions of Super Cereal Plus (SC+) 800 kcal per day associated with food ration for household support during hunger gap (5 months)
- Cash transfer: Monthly distributions of cash transfer only during hunger gap (5 months)

SUMMARY:
Options for large-scale preventive distributions include fortified blended flours, ready-to-use foods and direct cash transfer either alone or in combination with family protective rations. Finding the most appropriate strategy is essential to prevent child malnutrition in countries like Niger with annual hunger gaps. Here, the investigators compare different preventive strategies on the incidence of acute malnutrition among children 6 to 23 months.

ELIGIBILITY:
Inclusion Criteria:

* resident in selected villages
* height between 60 and 80 cm.

Exclusion Criteria:

* refusal to participate

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 6 to 24 months
Sampling Method: Non-Probability Sample
Enrollment: 7836 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Incidence of severe acute malnutrition | 15 months
  Severe acute malnutrition was defined as : Weight for Height Z-score (WHO Standards 2006)< -3 and/or mid-upper arm circumference (MUAC) < 115mm and/or bipedal oedema. MUAC was measured at the midpoint of a child's left arm with a plastic measuring tape with a precision of 1 mm.
  These indicators were evaluated monthly during the entire follow-up (15 months).

SECONDARY OUTCOMES:
Mortality | duration of follow-up (15 months)
  Mortality events include all reports for which the cause for absence from surveillance visits was reported to be death by a family member.

CONTACTS AND LOCATIONS:
Overall Officials: Céline Langendorf, MPH, Principal Investigator — Epicentre
Locations (1):
- Villages, Madarounfa, Maradi Region, Niger

REFERENCES:
- [Derived] Sayyad-Neerkorn J, Langendorf C, Roederer T, Doyon S, Mamaty AA, Woi-Messe L, Manzo ML, Harouna S, de Pee S, Grais RF. Preventive Effects of Long-Term Supplementation with 2 Nutritious Food Supplements in Young Children in Niger. J Nutr. 2015 Nov;145(11):2596-603. doi: 10.3945/jn.115.213157. Epub 2015 Sep 30. PMID 26423742
- [Derived] Langendorf C, Roederer T, de Pee S, Brown D, Doyon S, Mamaty AA, Toure LW, Manzo ML, Grais RF. Preventing acute malnutrition among young children in crises: a prospective intervention study in Niger. PLoS Med. 2014 Sep 2;11(9):e1001714. doi: 10.1371/journal.pmed.1001714. eCollection 2014 Sep. PMID 25180584